CLINICAL TRIAL: NCT06913348
Title: Ultrasound-Guided Sciatic Popliteal Nerve Block vs. Erector Spinae Plane Block in Patients Undergoing Endovascular Management of Critical Lower Limb Ischemia
Brief Title: Ultrasound-Guided Sciatic Popliteal Nerve Block vs. Erector Spinae Plane Block in Endovascular Management of CLI
Status: Completed | Type: Observational
Sponsor: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed hassan ahmed, Ultrasound guided sciatic popliteal nerve block versus Erector spinae plane block in patients undergoing endovascular management of critical lower limb ischemia., Minia University Hospital
Other Study IDs: ID number (1226/07/2024)
Record Dates: First submitted 2025-03-01; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Critical Limb Ischemia (CLI); Popliteal Nerve Block; ESPB
Keywords: popliteal nerve block; ESPB
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — comparison of popliteal sciatic nerve block versus ESPB .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ultrasound-Guided Sciatic Popliteal Nerve Block Group: Patients in this group will receive an ultrasound-guided sciatic popliteal nerve block for anesthesia during endovascular management of critical lower limb ischemia.
  Interventions: Procedure: Popliteal sciatic nerve block
- Erector Spinae Plane Block Group: Patients in this group will receive an ultrasound-guided erector spinae plane block for anesthesia during endovascular management of critical lower limb ischemia.
  Interventions: Procedure: Popliteal sciatic nerve block

INTERVENTIONS:
Procedure: Popliteal sciatic nerve block — Procedure/Surgery: Patients will receive either an ultrasound-guided sciatic popliteal nerve block or an ultrasound-guided erector spinae plane block for anesthesia during endovascular management of critical lower limb ischemia.

SUMMARY:
Comparison of popliteal sciatic nerve block and erector spinae plane block (ESPB) in patients undergoing endovascular management of critical lower limb ischemia (CLI).

DETAILED DESCRIPTION:
Nerve blocks, particularly regional anesthesia techniques, have been increasingly used in the endovascular management of critical lower limb ischemia (CLI). These techniques offer numerous advantages over general and local anesthesia.

Primary Advantages of Nerve Blocks:

1. Superior Pain Control

   Nerve blocks, such as femoral and sciatic nerve blocks, provide effective pain relief by anesthetizing the nerve supply to the lower limb.

   They offer more comprehensive analgesia than local anesthesia alone, as they numb the entire area around the puncture site.
2. Enhanced Patient Comfort

   Nerve blocks allow patients to remain pain-free during and after the procedure.

   They minimize discomfort even in lengthy or complex cases.
3. Reduction in Systemic Analgesic Requirements

   By providing localized anesthesia, nerve blocks significantly reduce the need for systemic analgesics, particularly opioids.

   This is essential because CLI patients often have comorbidities that make opioid use risky.
4. Fewer Opioid-Related Side Effects

   Nerve blocks reduce the incidence of opioid-related side effects, including nausea, vomiting, respiratory depression, and sedation.
5. Improved Hemodynamic Stability

Nerve blocks preserve autonomic nervous system function, reducing fluctuations in blood pressure and heart rate compared to general anesthesia.

This is especially beneficial for CLI patients, who frequently have underlying cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age will be 20-70 years.
2. Patients will be diagnosed with critical lower limb ischemia by clinical presentations and investigations.
3. ASA physical status 2-3

Exclusion Criteria:

1. Patient refusal to participate in this study.
2. Patient inability to understand the scales or to describe to the investigators.
3. Coagulation disorder.
4. Sever renal or kidney dysfunction.
5. Taking opioids before admission.
6. Morbid obesity .

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both sexes and from 20 to 80 years
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Block quality | Baseline (immediately after block administration).
  Assessment of the occurrence of complete motor and sensory block.

SECONDARY OUTCOMES:
Postoperative Analgesia Duration | Up to 24 hours postoperatively.
  Time from block administration to the first request for rescue analgesia.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Amr Nady Abd Elrazik, assistant professor, Study Director — Minia University Hospital
Locations (1):
- Minia university hospital, Minya, Minia Governorate, Egypt